CLINICAL TRIAL: NCT05817253
Title: Impact Evaluation of the Therapeutic Initiative's Uncomplicated Acute Cystitis Personalized Portrait and Therapeutics Letter
Brief Title: Evaluation of Therapeutic Initiative's Cystitis Portrait and Therapeutics Letter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Ministry of Health, British Columbia (Other Government)
Responsible Party: Principal Investigator, Colin Dormuth, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: H22-01140
Record Dates: First submitted 2023-02-09; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Clinical Audit; Quality Improvement
Keywords: Randomized Controlled Trial

STUDY DESIGN:
Intervention Model Description: Participants have been randomly divided into three groups which received the intervention at different times. Pooled data on the primary outcome (first-line prescribing for uncomplicated UTI) of those who received the intervention (mailed copy of personalized Portrait) early will be compared to that of those who received the delayed intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Letter + Portrait Arm (Experimental): Early Letter + Portrait Arm received a Portrait + Therapeutics Letter with the initial mailing (September 23, 2021). At the delayed mailing (March 28, 2022), Early Letter + Portrait Arm received nothing.
  Interventions: Behavioral: Portrait; Behavioral: Therapeutics Letter
- Delayed Control Arm (Experimental): Delayed Control Arm received nothing with the initial mailing (on September 23, 2021). At the delayed mailing (March 28, 2022), Delayed Control Arm received a Portrait +Therapeutics Letter.
  Interventions: Behavioral: Portrait; Behavioral: Therapeutics Letter
- Early Letter Arm (Experimental): Early Letter Arm received a Therapeutics Letter only with the initial mailing (September 23, 2021). At the delayed mailing (March 28, 2022), Early Letter Arm received a Portrait + Therapeutics Letter
  Interventions: Behavioral: Portrait; Behavioral: Therapeutics Letter

INTERVENTIONS:
Behavioral: Portrait — In the context of audit and feedback interventions, Portrait is document produced by the physician organization 'Therapeutics Initiative' that provides personalized prescribing feedback for BC family physicians (FPs). Portraits are used as a practice resource tool for reflection on prescribing patterns. Each Portrait topic provides data of individual physician's prescribing practice, alongside the mean and median levels of their peers (other BC physicians), a succinct review of the best-available evidence on the topic, and recommendations for future action.
Behavioral: Therapeutics Letter — The Therapeutics Letter is a standalone publication that details identified problematic therapeutic issues in a brief, simple and practical manner. Therapeutics letters include a systematic literature review on a clinical topic, and help provide reference for the data presented in the Portraits.

SUMMARY:
The goal of this randomized trial is to test the impact of mailing personalized prescribing Portraits (an audit and feedback tool) and Therapeutics Letters (a reference document) to physicians on first-line prescribing to patients with uncomplicated urinary tract infection (UTI) .

The main question this study aims to answer is:

• To what extent can personal prescribing feedback Portraits and Therapeutics Letters have an effect on how physicians prescribe antibiotics for uncomplicated UTI?

Approximately 5,000 British Columbian Family Practitioners (FP's) have been randomly divided into three groups, and each group received the Portrait at different times. To help ascertain the possible impact of Portraits, pooled data on first-line prescribing for uncomplicated UTI by FP's who received the Portrait at an early time point (September 23, 2021) will be compared to that of those who received a Portrait at a delayed time point (March 28, 2022). Researchers will compare prescribing data from these groups to see if the prescribing Portraits have had a differential impact on prescribing of antibiotics for uncomplicated UTI.

DETAILED DESCRIPTION:
This study is a randomized trial testing the effectiveness of personalized prescribing Portraits and Therapeutics Letters on appropriate treatment for uncomplicated acute cystitis (urinary tract infection) in the primary care setting in the province of British Columbia (B.C.) between September, 2021 and March, 2022.

Approximately 5,000 B.C. physicians were randomly divided into 3 arms (each representing ~ 33%) that received the Portrait and Therapeutics Letter at different times. Approximately 1,691 physicians were randomized to each group. This "designed delay" will enable evaluation of the impact of Portraits and Therapeutics Letters on prescribing at an aggregate level across the province of British Columbia.

On the initial mailing (September 23, 2021), Early Letter + Portrait Arm received a early Portrait (P) + Letter (L), Delayed Control Arm received nothing, and Early Letter Arm received an Early Letter Only. On the delayed mailing (March 28, 2022), both Early Letter Arm and Delayed Control Arm received a delayed Portrait (P) + Letter (L).

Within the study and across these groups, there will be four comparisons as follows:

During the study period (Sept 23, 2021 to Mar 28, 2022):

i. Early Letter + Portrait Arm vs Delayed Control Arm (to test the impact of L+P combined) ii. Early Letter + Portrait Arm vs Early Letter Arm (to test the the added impact of P in physicians who received L) iii. Early Letter Arm vs Delayed Control Arm (to test the the impact of L)

During the study period (Sept 23, 2021 to Sept 28, 2022):

iv. Delayed Control Arm vs Early Letter Arm (to test the impact of repeated messaging)

The analysis will identify:

1. Baseline Characteristics: Physicians and Patients by Study Group. Age (mean, sd), age groups, sex, urban vs rural.
2. Trends: monthly prescribing line chart for all of B.C. of Nitrofurantoin, Ciprofloxacin, and Trimethoprim-sulfamethoxazole (TMP-SMX), from 1 year prior to first mailing (September 23, 2021) to the end of the delay period (September 2022). This will illustrate background trends in prescribing patterns.
3. Relative Risk: Prescribing in the early and delayed intervention groups will be compared 6 months pre/post intervention. A four-way comparison of numerators during the pre/post periods between the early and delay groups will provide an odds ratio that approximates the relative risk.

ELIGIBILITY:
Inclusion Criteria:

Physicians who are:

i. Registered with the College of Physicians and Surgeons of B.C. (CPSBC) ii. Defined as a General Practitioner or Family Practice - Emergency Medicine according to the B.C. Ministry of Health's Medical Services Plan (MSP) with a license status of private practice, temporary license, salaried, or post graduate.

iii. Hold a valid mailing address in B.C according to the College of Physicians and Surgeons of British Columbia's public physician information.

iv. Had >=100 prescriptions filled at a community pharmacy in 2020 according to PharmaNet claims.

v. Diagnosed >= 1 eligible patient with Uncomplicated Acute Cystitis (UAC) in 2019 or 2020 (for delay group: 2020 to 2021

Exclusion Criteria:

Non-physicians, or physicians who:

i. Were not registered with the College of Physicians and Surgeons of B.C. (CPSBC) ii. Were not classified as a General Practitioner or Family Practice - Emergency Medicine according to the B.C. Ministry of Health's Medical Services Plan (MSP) with a license status of private practice, temporary license, salaried, or post graduate.

iii. Had an invalid mailing address in B.C according to the College of Physicians and Surgeons of British Columbia's public physician information.

iv. Had <=100 prescriptions filled at a community pharmacy in 2020 according to PharmaNet claims.

v. Diagnosed <= 1 eligible patient with Uncomplicated Acute Cystitis (UAC) in 2019 or 2020 (for delay group: 2020 to 2021

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5073 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Monthly prescribing of Nitrofurantoin | The study period for the primary analysis is the 185 day period after the early intervention, which is from September 24, 2021 to March 28, 2022..
  The primary outcome is the proportion of uncomplicated acute cystitis episodes treated with nitrofurantoin.

SECONDARY OUTCOMES:
Monthly prescribing of ciprofloxacin, trimethoprim-sulfamethoxazole (TMP-SMX), and other antibiotics. | The study period for the primary analysis is the 185 day period after the early intervention, which is from September 24, 2021 to March 28, 2022.
  Secondary outcomes are the proportion of uncomplicated acute cystitis episodes treated with ciprofloxacin, trimethoprim-sulfamethoxazole (TMP-SMX), and other antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Dormuth, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Therapeutics Initiative - Dept of Anesthesiology, Pharmacology & Therapeutics Faculty of Medicine University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Carney G, Maclure M, Patrick DM, Otte J, Ambasta A, Thompson W, Dormuth C. Pragmatic randomised trial assessing the impact of peer comparison and therapeutic recommendations, including repetition, on antibiotic prescribing patterns of family physicians across British Columbia for uncomplicated lower urinary tract infections. BMJ Qual Saf. 2025 Apr 17;34(5):295-304. doi: 10.1136/bmjqs-2024-017296. PMID 39414374

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT05817253/Prot_SAP_000.pdf